CLINICAL TRIAL: NCT04540211
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Study of Atezolizumab Plus Tiragolumab in Combination With Paclitaxel and Cisplatin Compared With Paclitaxel and Cisplatin as First-Line Treatment in Patients With Unresectable Locally Advanced, Unresectable Recurrent, or Metastatic Esophageal Squamous Cell Carcinoma
Brief Title: A Study of Atezolizumab Plus Tiragolumab in Combination With Paclitaxel and Cisplatin Compared With Paclitaxel and Cisplatin as First-Line Treatment in Participants With Unresectable Locally Advanced, Unresectable Recurrent, or Metastatic Esophageal Carcinoma
Acronym: SKYSCRAPER-08
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YO42138
Record Dates: First submitted 2020-09-03; First posted 2020-09-07 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — atezolizumab; Tiragolumab; Paclitaxel; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Atezolizumab + Tiragolumab + PC (Experimental): Participants will receive atezolizumab and tiragolumab on Day 1 of each 21-day cycle during the study followed by paclitaxel and cisplatin on Day 1 of each 21-day cycle until disease progression, loss of clinical benefit or unacceptable toxicity, during the induction treatment phase.
  Interventions: Drug: Atezolizumab; Drug: Tiragolumab; Drug: Paclitaxel; Drug: Cisplatin
- Placebo + PC (Placebo Comparator): Participants will receive atezolizumab matching placebo and tiragolumab matching placebo on Day 1 of each 21-day cycle during the study followed by paclitaxel and cisplatin on Day 1 of each 21-day cycle until disease progression, loss of clinical benefit or unacceptable toxicity, during the induction treatment phase.
  Interventions: Drug: Paclitaxel; Drug: Cisplatin; Drug: Atezolizumab Matching Placebo; Drug: Tiragolumab Matching Placebo

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab at a fixed dose of 1200 milligrams (mg) administered by intravenous (IV) infusion every 3 weeks (Q3W) on Day 1 of each 21-day cycle.
  Other Names: Tecentriq
  Arms: Atezolizumab + Tiragolumab + PC
Drug: Tiragolumab — Tiragolumab at a fixed dose of 600 mg administered by IV infusion every Q3W on Day 1 of each 21-day cycle.
  Other Names: MTIG7192A
  Arms: Atezolizumab + Tiragolumab + PC
Drug: Paclitaxel — Paclitaxel 175 mg/m^2 administered by IV infusion on Day 1 of each 21-day cycle for 6 cycles.
Drug: Cisplatin — Cisplatin 60-80 mg/m^2 administered by IV infusion on Day 1 of each 21-day cycle for 6 cycles.
Drug: Atezolizumab Matching Placebo — Atezolizumab matching placebo administered by IV infusion, Q3W on Day 1 of each 21-day cycle.
  Arms: Placebo + PC
Drug: Tiragolumab Matching Placebo — Tiragolumab matching placebo administered by IV infusion, Q3W on Day 1 of each 21-day cycle.
  Arms: Placebo + PC

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of atezolizumab plus tiragolumab in combination with paclitaxel and cisplatin (PC) compared with atezolizumab matching placebo plus tiragolumab matching placebo plus PC as first-line treatment in participants with unresectable locally advanced, unresectable recurrent, or metastatic esophageal carcinoma (EC). Participants will be randomized in a 1:1 ratio to receive one of the following treatment regimens during induction phase:

Arm A: Atezolizumab plus Tiragolumab and PC Arm B: Atezolizumab placebo plus Tiragolumab placebo and PC Following the induction phase, participants will continue maintenance therapy with either atezolizumab plus tiragolumab (Arm A) or atezolizumab matching placebo plus tiragolumab matching placebo (Arm B).

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed EC
* Unresectable locally advanced, unresectable recurrent, or metastatic disease
* Measurable disease per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1)
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Adequate hematologic and end-organ function
* Female participants must be willing to avoid pregnancy and refrain from donating eggs during the treatment period and for 90 days after the final dose
* Male participants with partners of childbearing potential must commit to the use of two methods of contraception and must not donate sperm for the study duration and 90 days after the final dose

Key Exclusion Criteria:

* Palliative radiation treatment for EC within 4 weeks prior to initiation of study treatment
* Evidence of complete esophageal obstruction not amenable to treatment
* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases
* Uncontrolled tumor-related pain, uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
* Active or history of autoimmune disease or immune deficiency or leptomeningeal disease
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis
* Malignancies other than EC within 2 years prior to screening with a negligible risk of metastasis or death adequately treated with expected curative outcome
* Severe infection within 4 weeks prior to initiation of study treatment or any active infection that, in the opinion of the investigator, could impact patient safety
* Positive test result for human immunodeficiency virus (HIV)
* Active hepatitis B or hepatitis C
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, anti-CTLA-4, anti-TIGIT, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* Treatment with any investigational therapy prior to initiation of study treatment
* Poor peripheral venous access
* Prior allogeneic stem cell or solid organ transplantation
* Concurrent participation in another therapeutic clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 461 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2025-08-28 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | From randomization to death from any cause (up to approximately 35 months)
Independent Review Facility (IRF)-Assessed Progression-Free Survival (PFS) | From randomization to the first occurrence of disease progression or death from any cause, whichever occurs first (up to approximately 35 months)

SECONDARY OUTCOMES:
Investigator-Assessed PFS | From randomization to the first occurrence of disease progression or death from any cause, whichever occurs first (up to approximately 35 months)
IRF-Assessed Confirmed Objective Response Rate (ORR) | From randomization up to approximately 35 months
Investigator-Assessed Confirmed ORR | From randomization up to approximately 35 months
IRF-Assessed Duration of Objective Response (DOR) | From the first occurrence of a documented confirmed objective response to the first occurrence of disease progression or death from any cause, whichever occurs first (up to approximately 35 months)
Investigator-Assessed DOR | From the first occurrence of a documented confirmed objective response to the first occurrence of disease progression or death from any cause, whichever occurs first (up to approximately 35 months)
Time to Confirmed Deterioration (TTCD) in Participant-Reported Physical Functioning, Role Functioning and Global Health Status (GHS)/Quality of Life (QoL) as Measured by EORTC QLQ-C30 | From randomization until the first confirmed clinically meaningful deterioration (up to approximately 35 months)
  Clinically meaningful changes in physical functioning, role functioning, global health status (GHS)/QoL as measured by the European Organisation for Research and Treatment of Cancer Quality of Life-Core 30 Questionnaire (EORTC QLQ-C30). EORTC QLQ-C30 is a self-reported measure, consisting of 30 questions that assess 5 aspects of participants functioning (physical, emotional, role, cognitive and social), 3 symptom scales (fatigue, nausea and vomiting, and pain), GHS and QoL, and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties) within the previous week. Functioning and symptoms items are scored on a 4-point scale: 1=Not at all, 2=A little, 3=Quite a bit, 4=Very much. GHS and QoL items are scored on a 7-point scale: 1=Very poor, 2, 3, 4, 5, 6, 7=Excellent. Scores will be linearly transformed to a range of 0 to 100, with higher scores (i.e. closer to 100) reflecting better functioning, better GHS/QoL, and worse symptoms.
TTCD in Participant-Reported Dysphagia as Measured by EORTC QLQ-OES18 | From randomization until the first confirmed clinically meaningful deterioration (up to approximately 35 months)
  Clinically meaningful changes in dysphagia as measured by the EORTC Quality of Life-Esophageal Cancer, Module 18 Questionnaire (EORTC QLQ-OES18). EORTC QLQ-OES18 is a modular supplement to the EORTC QLQ-C30 questionnaire for use in participants with esophageal cancer. EORTC QLQ-OES18 consists of 4 multiple-item scale (dysphagia, eating, reflux, and pain) and 6 single items (trouble swallowing saliva, choked when swallowing, dry mouth, trouble with taste, trouble with coughing, and trouble talking) with a recall period of the previous week. Each symptom item is scored on a 4-point scale: 1=Not at all, 2=A little, 3=Quite a bit, 4=Very much. Scores will be linearly transformed to a range of 0 to 100, with higher transformed scores (i.e. closer to 100) reflecting worse symptoms.
Percentage of Participants With Adverse Events (AEs) | Up to approximately 35 months
Minimum Serum Concentration (Cmin) of Tiragolumab | Cycle 1 (cycle=21 days), Day 1: predose, 0.5 hour (h) postdose; Cycles 2, 3, 4, 8, 12, 16, Day 1: predose and at treatment discontinuation (TD) visit (up to approximately 35 months)
Maximum Serum Concentration (Cmax) of Tiragolumab | Cycle 1 (cycle=21 days), Day 1: predose, 0.5h postdose; Cycles 2, 3, 4, 8, 12, 16: Day 1: predose and at TD visit (up to approximately 35 months)
Cmin of Atezolizumab | Cycle 1 (cycle=21 days): Day 1 (predose, 0.5 h postdose); Cycles 2, 3, 4, 8, 12, 16: Day 1 (predose) and at TD visit (up to approximately 35 months)
Cmax of Atezolizumab | Cycle 1 (cycle=21 days): Day 1 (predose, 0.5 h postdose); Cycles 2, 3, 4, 8, 12, 16: Day 1 (predose) and at TD visit (up to approximately 35 months)
Percentage of Participants With Anti-drug Antibodies (ADAs) to Tiragolumab | Predose on Day 1 of Cycles (cycle=21 days) 1, 2, 3, 4, 8, 12 and 16 and at TD visit (up to approximately 35 months)
Percentage of Participants With ADAs to Atezolizumab | Predose on Day 1 of Cycles (cycle=21 days) 1, 2, 3, 4, 8, 12 and 16 and at TD visit (up to approximately 35 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (64):
- China (46):
  - Anhui Provincial Hospital, Anhui
  - Anyang Tumor Hosptial, Anyang
  - Beijing Cancer Hospital, Beijing
  - Beijing Luhe Hospital Capital Medical University, Beijing
  - Jilin Cancer Hospital, Changchun
  - Hunan Cancer Hospital, Changsha
  - Affiliated Hospital of Chengde Medical University, Chengde
  - Sichuan Provincial Cancer Hospital, Chengdu
  - West China Hospital, Sichuan University, Chengdu
  - Chongqing Sanxia Central Hospital, Chongqing
  - Fujian Cancer Hospital, Fuzhou
  - Fujian Provincial Hospital, Fuzhou
  - Southern Medical University Nanfang Hospital, Guangdong Province Guangzhou City
  - Zhejiang Cancer Hospital, Hangzhou
  - Anhui Province Cancer Hospital, Hefei
  - The Second Affiliated Hospital of Anhui Medical University, Hefei
  - Huai'an First People's Hospital, Huai'an
  - The Second People's Hospital of Huai'an, Huai'an
  - Affiliated Hopsital of Jining Medical University, Jining
  - Gansu Province People Hospital, Lanzhou
  - The First People's Hospital of Lian Yun Gang, Lianyungang
  - Linyishi Cancer Hospital, Linyi
  - Jiangsu Province Hospital of Chinese Medicine, Nanjing
  - Jiangsu Cancer Hospital, Nanjing
  - Nan Tong Tumor Hospital, Nantong
  - Shanghai Chest Hospital, Shanghai
  - Zhongshan Hospital Fudan University, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Cancer Hospital of Shantou University Medical College, Shantou
  - Liaoning Provincial Cancer Hospital, Shengyang
  - Suining Central Hospital, Suining
  - Tianjin Cancer Hospital, Tianjin
  - Weifang People's Hospital, Weifang
  - Wuhan Union Hospital Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Hubei Cancer Hospital, Wuhan
  - Affiliated Hospital of Jiangnan University(Wuxi Fourth People's Hospital ), Wuxi
  - The Second Affiliated Hospital of The Fourth Military Medical University (Tangdu Hospital), Xi'an
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi'an
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Zhongshan Hospital Xiamen University, Xiamen
  - Xiangyang Central Hospital, Xiangyang
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang
  - Xuzhou Central Hospital, Xuzhou
  - Northern Jangsu People's Hospital, Yangzhou
  - Henan Cancer Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hosp, Shatin
- South Korea (7):
  - Kyungpook National University Chilgok Hospital, Daegu
  - National Cancer Center, Goyang-si
  - Seoul National University Bundang Hospital, Seongnam-si
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
- Taiwan (4):
  - Chang Gung Medical Foundation - Kaohsiung, Kaohisung
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
  - National Taiwan University Hospital, Zhongzheng Dist.
- Thailand (5):
  - Chulalongkorn Hospital, Bangkok
  - Rajavithi Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Songklanagarind Hospital, Songkhla

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Sun JM, Chao Y, Kim SB, Rha SY, Evans TRJ, Strickland AH, Wainberg Z, Chau I, Pelles-Avraham S, Ajani J, Malhotra R, Liu Q, Li S, Cha E, Kalaitzidou M, Huang X, Allen S, Hsu CH. First-line tiragolumab plus atezolizumab and chemotherapy in patients with previously untreated, locally advanced unresectable or metastatic oesophageal cancer (MORPHEUS-EC): a randomised, open-label, phase 1b/2 trial. Lancet Oncol. 2026 Jan;27(1):90-102. doi: 10.1016/S1470-2045(25)00402-4. PMID 41449151
- [Derived] Hsu CH, Lu Z, Gao S, Wang J, Sun JM, Liu T, Fan Q, Cai J, Ge F, Li S, Zhang L, Cha E, Allen S, Shen L. Tiragolumab plus atezolizumab and chemotherapy as first-line treatment for patients with unresectable oesophageal squamous cell carcinoma (SKYSCRAPER-08): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2026 Jan;27(1):103-115. doi: 10.1016/S1470-2045(25)00401-2. PMID 41449142